CLINICAL TRIAL: NCT01148498
Title: Plasma Amyloid Beta Species After a Single Solanezumab Infusion in Nondemented Individuals and Those With Mild Dementia of the Alzheimer's Type
Brief Title: A Biomarker Study of Solanezumab in Patients With and Without Alzheimer's
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13572; H8A-MC-LZAT (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — solanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): Older adults with mild Dementia Alzheimer's Type (DAT)
  Interventions: Drug: solanezumab
- Group 2 (Experimental): Older adult controls with possible Alzheimer's Disease Pathology
  Interventions: Drug: solanezumab
- Group 3 (Experimental): Older adult controls with no evidence of Alzheimer's Disease
  Interventions: Drug: solanezumab
- Group 4 (Experimental): Younger subjects who are assumed to have no cognitive impairment
  Interventions: Drug: solanezumab

INTERVENTIONS:
Drug: solanezumab — 400mg administered once intravenously
  Other Names: LY2062430; A Beta Antibody

SUMMARY:
The purpose of this trial is to compare the average change in the amount of amyloid beta species in blood after an infusion of solanezumab.

ELIGIBILITY:
Inclusion Criteria:

Individuals in Groups 1, 2, and 3, described below, will be participants in the longitudinal studies of memory and aging at the Washington University Alzheimer's Disease Research Center (WU-ADRC). These participants must have results from apolipoprotein E (ApoE) genotyping from the WU-ADRC. At the beginning of the study they must be between 45 and 90 years of age and if a female of childbearing potential, not be breastfeeding, test negative for pregnancy, and be using a medically accepted form of birth control at the time of the infusion and for 6 months afterward. Subjects must also meet the criteria below for each study group

Group 1, Mild dementia of Alzheimer's type (DAT):

* Have mild DAT, as determined by Clinical Dementia Rating (CDR) of 0.5 or 1
* Have florbetapir PET imaging findings consistent with underlying AD pathology.

Group 2, Older Adult Controls with Possible AD Pathology:

Have no cognitive impairment as indicated by a CDR rating of 0. Have possible AD pathology, as determined by florbetapir PET imaging.

Group 3, Older Adult Controls with No Evidence of AD Pathology:

Have no cognitive impairment as indicated by a CDR rating of 0. Have no evidence of AD pathology as determined by florbetapir PET imaging.

Individuals recruited into Group 4 will not be participants in the longitudinal studies of memory and aging at WU-ADRC. To be included in Group 4, individuals must meet these criteria:

* Are at least 18 years and <35 years of age at the beginning of the study and if a female of childbearing potential, is not breastfeeding, tests negative for pregnancy and is using highly effective contraception at the time of the solanezumab infusion and for 6 months following infusion
* Have a Folstein Mini-Mental State Examination (MMSE) score of 29 to 30 at the beginning of the study

Exclusion Criteria:

* Have previously completed or withdrawn from this study or any other study investigating solanezumab
* Does not have good venous access, such that intravenous drug delivery or multiple blood draws would be precluded
* Has allergies to humanized monoclonal antibodies
* Has a known history of human immunodeficiency virus (HIV), clinically significant multiple or severe drug allergies, or severe posttreatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear IgA dermatosis, toxic epidermal necrolysis, or exfoliative dermatitis)
* Has a history of chronic alcohol or drug abuse/dependence
* Is clinically judged by the investigator to be at serious risk for suicide
* Has a recent (within 6 months before screening) or current laboratory result (if available) indicating a clinically significant laboratory abnormality
* Has Electrocardiogram (ECG) abnormalities obtained at screening that, in the opinion of the investigator, are clinically significant with regard to the subject's participation in the study. Bazett's corrected QT [QTcB] interval must be evaluated and must not exceed >458 msec in males or >474 msec in females
* At screening, has alanine transaminase (ALT/SGPT) values greater than or equal to 2 times the upper limit of normal (ULN) of the performing laboratory, aspartate transaminase (AST/SGOT) values greater than or equal to 3 times the ULN, or total bilirubin values greater than or equal to 2 times the ULN
* Has had IgG therapy (sometimes called gamma globulin therapy) within the last year or previous participation in any other study investigating active immunization against Aβ
* Requires treatment with other monoclonal antibodies

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline up to 112 days post drug administration in plasma levels of Aβ fragment-2 in (Group 1) and (Group 3) | Baseline up to 112 days post drug administration

SECONDARY OUTCOMES:
Mean change in plasma levels of Aβ1-42 after solanezumab infusion | Baseline (pre-dose); 30 minutes; 24 hours; 7, 28, 56 and 112 days post-dose
Mean change in plasma levels of Aβ1-40 species after solanezumab infusion | Baseline (pre-dose); 30 minutes; 24 hours; 7, 28, 56 and 112 days post-dose
Mean change in plasma levels of modified Aβ species after solanezumab infusion | Baseline (pre-dose); 30 minutes; 24 hours; 7, 28, 56 and 112 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri, United States